CLINICAL TRIAL: NCT07222995
Title: A Hybrid Effectiveness-Implementation Trial to Integrate Precision Skin Cancer Risk Feedback in Federal Qualified Health Centers
Brief Title: Hybrid Effectiveness-Implementation Trial to Integrate Precision Skin Cancer Risk Feedback in FQHCs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-23436
Record Dates: First submitted 2025-10-28; First posted 2025-10-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Precision Prevention Intervention (Active Comparator): Participants receive personalized skin cancer prevention materials based on MC1R genetic risk.
  Interventions: Behavioral: Precision Prevention Booklet
- Standard Prevention (Active Comparator): Participants receive standard skin cancer prevention materials.
  Interventions: Behavioral: Standard Prevention Booklet
- Non-Intervention (No Intervention): Participants who do not return saliva kits will not receive intervention materials but will complete follow-up assessments.

INTERVENTIONS:
Behavioral: Precision Prevention Booklet — Precision prevention booklet anchored in their MC1R risk that incorporates gold-standard risk communication strategies, including visual risk representations and simple language.
  Arms: Precision Prevention Intervention
Behavioral: Standard Prevention Booklet — Standard materials are similar in content to the precision prevention booklet but without any reference to MC1R risk.
  Arms: Standard Prevention

SUMMARY:
The purpose of this study is to examine how different messages about risk of skin cancer can impact the uptake of skin cancer prevention activities.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient of any race or ethnicity attending one of the six Tampa Family Health Centers.
* Be 18 years of age or older.
* Self-report skin cancer risk behaviors within the past 12 months, including: Intentional sun exposure (e.g., outdoor or indoor tanning) or unintentional sun exposure leading to sunburn.
* Be willing to complete a baseline questionnaire and provide a saliva sample for MC1R genotyping.
* Be able to provide informed consent (written or electronic).
* Prefer English or Spanish for communication and study materials.

Exclusion Criteria:

* Do not report any skin cancer risk behaviors (i.e., no tanning or sunburning in the past 12 months).
* Are unwilling or unable to complete the baseline assessment or return the saliva kit.
* Decline to provide informed consent.
* Are under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2900 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2030-10-10 (Estimated); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in Tanning Score | Baseline, 6 months, 12 months
  Change in self-reported tanning behavior score from baseline to 6 and 12 months.
Number of Sunburns | Baseline, 6 months, 12 months
  Change in self-reported number of sunburns experienced over the past 6 and 12 months.
Skin self-examination (SSE) | Baseline, 6 months, 12 months
  Change in self-reported SSE from baseline to 6 and 12 months.
Physician-patient communication about skin cancer prevention. | Baseline, 6 months, 12 months
  Change in self-reported physician-patient communication from baseline to 6 and 12 months.

SECONDARY OUTCOMES:
Change in Hours Spent Outside in the Sun | Baseline, 6 months, 12 months
  Change in self-reported average weekly hours spent outdoors in direct sunlight, assessed via questionnaire.
Change in Sun Protection Behaviors | Baseline, 6 months, 12 months
  Change in frequency of sun protection behaviors, including use of sunscreen, wearing protective clothing, and seeking shade, assessed via a composite behavior scale.
Receipt of Total Body Skin Examination (TBSE) | 12 months
  Proportion of participants who report referral for and receiving a total body skin examination by a healthcare professional during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kanetsky, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York